CLINICAL TRIAL: NCT05419856
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Doses of 4P004 Versus Placebo Injected in the Target Knee of Patients With Grade 2 to 4 Osteoarthritis on the Kellgren and Lawrence Severity Index
Brief Title: Safety, Tolerability and Pharmacokinetics of Intraarticular 4P004 Single Dose in Patient With KL 2-4 Osteoarthritic Knee
Acronym: LASARE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 4Moving Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 4MB-LAS-P
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
Keywords: OA; Knee OA; Liraglutide
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: A total of 32 participants will be enrolled in 4 cohorts, in each cohort participants will receive either 4P-004 or placebo (6:2).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 4P-004 w mg (Experimental): 4P-004 is administered once intraarticularly in the target knee joint Dose = w mg
  Interventions: Drug: 4P-004
- 4P-004 x mg (Experimental): 4P-004 is administered once intraarticularly in the target knee joint Dose = x mg
  Interventions: Drug: 4P-004
- 4P-004 y mg (Experimental): 4P-004 is administered once intraarticularly in the target knee joint Dose = y mg
  Interventions: Drug: 4P-004
- 4P-004 z mg (Experimental): 4P-004 is administered once intraarticularly in the target knee joint Dose = z mg
  Interventions: Drug: 4P-004
- Placebo (Placebo Comparator): Placebo is administered once intraarticularly in the target knee joint
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4P-004 — single intraarticular administration in the knee joint
  Other Names: Liraglutide
  Arms: 4P-004 w mg; 4P-004 x mg; 4P-004 y mg; 4P-004 z mg
Drug: Placebo — single intraarticular administration in the knee joint
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
This phase I study is a multicenter, randomized, double-blind, placebo-controlled study to assess the safety and tolerability of single ascending dose of IA 4P-004 in participants,

* Between 18 and 80 years of age,
* with target knee OA stage KL 2-4 A total of 32 participants will be enrolled in 4 cohorts, in each cohort participants will receive either 4P-004 or placebo (6:2).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have the capacity to give informed consent and who are willing to comply with all study related procedures and assessments (consent via legally authorized representative will not be accepted),
* Ambulatory participants, agreeing a 24-hour hospitalization,
* Participants between 18 and 80 years of age,
* Female participant of childbearing potential (WOCBP), must use contraceptive consistent with local regulations regarding the methods of contraception for those participating in clinical studies (see section 11.4) for at least 5 days following IMP injection, and must have a negative urine pregnancy test done within 24h before randomization,
* Male participants (whose partners are of childbearing potential) must consent to use methods of contraception consistent with local regulations regarding the methods of contraception for those participating in clinical studies (see section 11.4), for at least 90 days following IMP injection,
* Participants with knee osteoarthritis, KL 2-4 of their target knee (defined at screening as the knee with greater pain based on the participant's evaluation and the investigator's clinical judgment),
* X-rays of the target knee within 6 months (if not, to be performed before randomization),
* ECG within normal range,
* WBC (white blood cell count) > 3500/µL,
* Hemoglobin > 12 g/dL,
* Platelets > 100,000/ µL,
* Creatinine clearance (CrCl) > 60 mL/min,
* Glycemia within normal range,
* AST, ALT < 1.5 upper limit of normal (ULN),
* Amylasemia < 1ULN,
* Negative tests for COVID-19 (if required by the standard practice on site), HIV, HbsAg and hepatitis C Ab (Determination of HIV and hepatitis status can be based on participant-reported medical history, available medical records, and the most recently available laboratory results for the participant [tests performed within the previous 12 months]).

Exclusion Criteria:

* Breastfeeding women,
* Treatment with systemic glucocorticoids greater than 10 mg prednisone or the equivalent per day within 4 weeks prior to screening,
* Any treatment with glucosamine or chondroitin sulfate in the previous 3 months,
* Any glucagon-like peptide 1 analogue hormones,
* Anticoagulant treatment (current or within the last 10 days),
* Treatment of the target knee with any IA injection (steroids, hyaluronic acid derivatives, PRP ….) within 3 months,
* Knee surgery (of the target knee) performed within the previous 12 months or planned within the next 6 months,
* Any partial knee replacement of the target knee,
* Any known active infections or increased predisposition for the development of infections
* Clinical signs and symptoms of active joint crystal disease, or any inflammatory joint disease,
* Diabetes type I or II,
* Congestive Heart Failure stage III or IV of NYHA classification,
* Inflammatory bowel disease,
* Any other chronic condition that has not been well controlled for a minimum of 3 months,
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer) within the last 5 years,
* Any condition, including laboratory findings, that in the opinion of the investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation, (for example, any abnormal reaction to previous IA injection),
* Hypersensitivity to the active substance liraglutide or to any of the excipients: Disodium phosphate dihydrate, Propylene glycol, Phenol,
* Participation in an interventional clinical research trial within 12 weeks prior.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - UCL-St Luc, Brussels
  - AZMaria Middelares, Ghent
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meurot C, Martin C, Sudre L, Breton J, Bougault C, Rattenbach R, Bismuth K, Jacques C, Berenbaum F. Liraglutide, a glucagon-like peptide 1 receptor agonist, exerts analgesic, anti-inflammatory and anti-degradative actions in osteoarthritis. Sci Rep. 2022 Jan 28;12(1):1567. doi: 10.1038/s41598-022-05323-7. PMID 35091584
- See also: 4Moving Biotech (sponsor) web site — https://www.4movingbiotech.com

RESULTS

PARTICIPANT FLOW:
Period: Cohort 1
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo
Started | 6 | 0 | 0 | 0 | 2
Completed | 6 | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 2
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo
Started | 0 | 6 | 0 | 0 | 2
Completed | 0 | 6 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 3
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo
Started | 0 | 0 | 6 | 0 | 2
Completed | 0 | 0 | 6 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 4
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo
Started | 0 | 0 | 0 | 8 | 2
Completed | 0 | 0 | 0 | 8 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 4P-004 w mg: 4P-004: single intraarticular administration in the knee joint Dose = w mg
- 4P-004 x mg: 4P-004: single intraarticular administration in the knee joint Dose = x mg
- 4P-004 y mg: 4P-004: single intraarticular administration in the knee joint Dose = y mg
- 4P-004 z mg: 4P-004: single intraarticular administration in the knee joint Dose = z mg
- Total: Total of all reporting groups
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (6.9) | 54.2 (5.3) | 60.3 (8.5) | 59.1 (59.5) | 63.5 (11.5) | 60.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 5 | 5 | 19
  Male | 3 | 4 | 2 | 3 | 3 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 29 (6.8) | 28 (5.1) | 28.5 (4.9) | 25.5 (5) | 29.5 (4.3) | 28.1 (5.1)
Kellgren-Lawrence score [Count of Participants; unit: Participants] — The KL classification is based on radiography assessment. Each radiograph was assigned a grade from 0 to 4, which they correlated to increasing severity of OA, with Grade 0 signifying no presence of OA and Grade 4 signifying severe OA
  Participants
    Kellgren-Lawrence 2 | 2 | 4 | 3 | 6 | 6 | 21
    Kellgren-Lawrence 3 | 4 | 1 | 3 | 1 | 2 | 11
    Kellgren-Lawrence 4 | 0 | 1 | 0 | 1 | 0 | 2
NRS [Mean (Standard Deviation); unit: units on a scale] — The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
  units on a scale | 3.8 (2.3) | 4.0 (2.0) | 3.5 (2.6) | 3.5 (2.3) | 3.7 (2.4) | 3.7 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Single IA Administration of 4P-004 at Escalating Doses in Participants With Knee OA.
Description: Number of participants with Adverse Events, serious AEs (SAEs), with abnormal Vital signs, abnormal ECG reading and abnormal Laboratory test results
Time Frame: Day 1-Day 28
Measure: Number; unit: participants
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 8
participants
  TEAE | 5 | 5 | 5 | 6 | 6
  SAE | 0 | 0 | 1 | 0 | 0
  Abnormal Vital Sign | 0 | 0 | 0 | 0 | 0
  Abnormal Laboratory Value | 0 | 0 | 0 | 0 | 0
  Abnormal ECG | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: To Characterize the Plasma Concentration of Liraglutide When Administered as Single IA Doses at Escalating Dose Levels in Participants With Knee OA
Description: Plasma concentration of liraglutide following a single IA injection at pre-injection (Time [-4hours-0]) and 2hours, 4hours, 8hours, 12hours, 16hours and 24-hours post injection.
Time Frame: Day 1 to Day 2
Population: Placebo participant where not included in the PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 7 | 0
ng/mL
  Time [-4hours-0] | 0 (0) | 0 (0) | 0 (0) | 0 (0) |
  Time 2 hours | 3.6 (1.1) | 7.2 (4.2) | 58.1 (38.8) | 24.6 (15.7) |
  Time 4 hours | 5.3 (1.8) | 13.9 (7.5) | 90.4 (58.6) | 41.6 (18.4) |
  Time 8 hours | 7.3 (3.1) | 23.2 (12.4) | 123.7 (74.9) | 64.5 (23.0) |
  Time 12 hours | 7.1 (3.1) | 24.5 (12.9) | 122.2 (69.2) | 67.2 (24.7) |
  Time 16 hours | 6.4 (2.9) | 23.5 (12.0) | 113.6 (61.8) | 63.8 (25.4) |
  Time 24 hours | 5.0 (2.4) | 20.0 (9.4) | 95.2 (52.1) | 53.6 (25.4) |

3. Other Pre Specified Outcome: Exploratory Biomarkers Identification
Description: Serum and urine OA-related biomarkers (exploratory proteomic research of 4P-004 efficacy-related biomarkers) at Day 1 (Time [-4-0]hours, Time 8hours), Day 2 (Time 24hours) and Day 8.
Time Frame: Day 1, Day 2, Day 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were collected from screening until the End of study (D29)
Arm/Group | 4P-004 w mg | 4P-004 x mg | 4P-004 y mg | 4P-004 z mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 5/6 | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4P-004 w mg (N=6) | 4P-004 x mg (N=6) | 4P-004 y mg (N=6) | 4P-004 z mg (N=8) | Placebo (N=8)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4P-004 w mg (N=6) | 4P-004 x mg (N=6) | 4P-004 y mg (N=6) | 4P-004 z mg (N=8) | Placebo (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 5 (8) | 2 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (2) | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 (2) | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 1 (1) | 2 (3) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 0 | 0 | 2 (3) | 1 (1) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 (2) | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 1 (2) | 2 (4) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 (1) | 1 (1) | 0 | 1 (1)
Injection site pain (General disorders) | 0 | 2 (2) | 0 | 0 | 0
Chest pain (General disorders) | 1 (1) | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 1 (1) | 0 | 0
Injection site joint pain (General disorders) | 0 | 0 | 0 | 1 (1) | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 | 1 (1) | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 1 (1) | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0
Hot flush (Vascular disorders) | 1 (1) | 0 | 0 | 0 | 1 (1)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The INSTITUTION and the INVESTIGATOR may not use any information other than publicly available information regarding the Study in any publicity and advertising without SPONSOR's prior written consent and ethics committee approval.

DOCUMENTS (2):
  • Study Protocol (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT05419856/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT05419856/SAP_001.pdf